CLINICAL TRIAL: NCT00282022
Title: A Phase II Trial of Cloretazine™ (VNP40101M) for Patients With Relapsed or Refractory Small Cell Lung Cancer
Brief Title: VNP40101M in Treating Patients With Relapsed or Refractory Locally Advanced or Metastatic Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456623; VION-CLI-039
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2009-01

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer; extensive stage small cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — laromustine

INTERVENTIONS:
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as VNP40101M, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well VNP40101M works in treating patients with recurrent or refractory locally advanced or metastatic small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate (partial and complete) in patients with relapsed or refractory locally advanced or metastatic small cell lung cancer treated with VNP40101M.
* Determine the toxic effects of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease state (sensitive relapse [progressive disease > 3 months after responding to first-line chemotherapy] vs resistant disease [progressive disease during or ≤ 3 months after first-line chemotherapy]).

Patients receive VNP40101M IV over 15-30 minutes once weekly for 3 weeks. Treatment repeats every 6 weeks for up to 6 courses. Patients achieving a complete response (CR) receive 2 additional courses of therapy after CR.

After completion of study treatment, patients are followed periodically for up to 18 months.

PROJECTED ACCRUAL: A total of 87 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed small cell lung cancer

  * Locally advanced or metastatic disease
  * Recurrent or progressive disease after first-line standard cytotoxic therapy
* Measurable or evaluable disease
* Brain metastasis allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 2 months
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.5 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled bleeding
* No active infection
* Must not require supplemental oxygen at rest
* No active heart disease
* No myocardial infarction within the past 3 months
* No uncontrolled congestive heart failure
* No uncontrolled arrhythmias
* No uncontrolled coronary artery disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior radiotherapy, biologic therapy or chemotherapy (6 weeks for nitrosoureas or mitomycin C)

  * Prior radiotherapy within the past 3 weeks allowed if exposure involves no more than 30% of bones with significant bone marrow-producing capabilities (e.g., vertebral bodies and long bones)
* At least 2 weeks since prior surgery or hormonal therapy
* Must not require any immediate palliative treatment including surgery
* Must have recovered from prior anticancer therapy

  * Persistent, stable chronic toxic effects ≤ grade 1 are allowed
* No more than 1 prior systemic chemotherapy regimen for locally advanced or metastatic disease
* No other concurrent anticancer therapy
* No other concurrent investigational agent
* No concurrent disulfiram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete and partial response)
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bonny L. Johnson, RN, MSN — Vion Pharmaceuticals
Locations (9):
- United States (9):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Veterans Affairs Medical Center - West Haven, West Haven, Connecticut
  - Helen F. Graham Cancer Center at Christiana Hospital, Newark, Delaware
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas